CLINICAL TRIAL: NCT07346027
Title: A Randomized, Open Labeled, Two-period, Two-sequence Crossover, Phase 1 Study of F-02-2-Na Tablets in Healthy Adult Subjects：Assessment of Food Effect on Single-Dose Bioavailability
Brief Title: Safety and Food Effect on Single-Dose Bioavailability of F-02-2-Na in Healthy Adult Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Hengqin Novagains Biopharmaceutical Co., Ltd. (Industry)
Collaborators: Xiangbei Welman Pharmaceutical Co., Ltd (Industry); Guangzhou Xin-Chuangyi Biopharmaceutical Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: F-02-2-Na-2025-PROT-I-2
Record Dates: First submitted 2025-11-28; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Hyperuricemia With or Without Gout

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FE-1 Fasting-Fed Group (Experimental): Fasting administration of F-02-2-Na - Fed administration of F-02-2-Na
  Interventions: Drug: Fasting administration of F-02-2-Na (50mg) - Fed administration of F-02-2-Na (50mg)
- FE-2 Fed-Fasting Group (Experimental): Fed administration of F-02-2-Na - Fasting administration of F-02-2-Na
  Interventions: Drug: Fed administration of F-02-2-Na (50mg) - Fasting administration of F-02-2-Na (50mg)

INTERVENTIONS:
Drug: Fasting administration of F-02-2-Na (50mg) - Fed administration of F-02-2-Na (50mg) — Firstly, subjects will receive a fasting administration of F-02-2-Na (50 mg); secondly, a washout period of at least 4 days will be implemented; thirdly, subjects will receive a fed administration of F-02-2-Na (50 mg).
  Other Names: FE-1 Fasting-Fed Group
  Arms: FE-1 Fasting-Fed Group
Drug: Fed administration of F-02-2-Na (50mg) - Fasting administration of F-02-2-Na (50mg) — Firstly, subjects will receive a fed administration of F-02-2-Na (50 mg); secondly, a washout period of at least 4 days will be implemented; thirdly, subjects will receive a fasting administration of F-02-2-Na (50 mg).
  Other Names: FE-2 Fed-Fasting Group
  Arms: FE-2 Fed-Fasting Group

SUMMARY:
The study is to evaluate the impact of food on the pharmacokinetics of F-02-2-Na in healthy adult subjects by observing the changes in the drug's pharmacokinetic profile-particularly in its absorption process-before and after food intake.

DETAILED DESCRIPTION:
Approximately 12 subjects will be enrolled in Food Effect clinical trial to conduct an open-label, 2-way crossover treatment study with follow-up period. Twelve subjects will be randomized just prior to dosing to one of the 2 treatment sequences according to a randomization schedule: Sequence 1 is Period 1 Fasted State-Washout -Period 2 Fed State; Sequence 2 is Period 1 Fed State-Washout-Period 2- Fasted State.

ELIGIBILITY:
Inclusion Criteria:

* 1. The subjects should fully understand the purpose, nature, process of the study and the possible adverse reactions, voluntarily act as subjects, and sign the informed consent form before the start of any research procedures.
* 2. Healthy male or female subjects aged 18 to 45 years old (inclusive).
* 3. The body weight for male and female subjects should be ≥ 50.0 kg and ≥ 45.0 kg, respectively; the body mass index (BMI) should be between 19 kg/m² and 26 kg/m² (inclusive).
* 4. The subjects should have normal results or abnormal results without clinical significance in vital signs check, physical examination, clinical laboratory tests (Complete Blood Count (CBC), urine analysis, blood biochemistry, coagulation panel, free thyroid function tests), chest X-ray, liver and renal color ultrasound and 12-lead electrocardiogram.
* 5. Normal renal function as determined by Investigator following review of clinical laboratory test results, including eGFR ≥ 90 mL/min/1.73 m².
* 6. The subjects (including male subjects) should have no plans for having children from screening until 6 months after the last dose and should voluntarily take effective contraceptive measures and have no plans for sperm or egg donation.
* 7. The subjects should be able to communicate well with the researchers and understand and comply with the requirements of this study.

Exclusion Criteria:

* 1. Subjects with a specific allergic history (such as asthma, urticaria, eczema, etc.) or those with an allergic constitution (such as those known to be allergic to two or more substances), or those with a known history of allergy to F-02-2-Na and related excipients (ascertained through inquiry).
* 2. Subjects who have had an acute illness within two weeks before the first drug administration (ascertained through inquiry).
* 3. Subjects with diseases of important organs or systems (including but not limited to liver, kidney, nervous system, blood, endocrine system, lungs, immune system, mental health, cardiovascular and cerebrovascular system, gastrointestinal tract, skin, metabolism, bone and joints, etc.) that are considered clinically significant by the researcher, or those with a history of such serious diseases; or those with a history of tumor (ascertained through inquiry).
* 4. Subjects with a history of gastrointestinal, liver, kidney, and thyroid diseases that can affect drug absorption or metabolism (ascertained through inquiry).
* 5. Subjects with a history of gout (ascertained through inquiry).
* 6. Subjects who have used any medications (including any prescription drugs, over-the-counter drugs, traditional Chinese herbal medicines) and health products within two weeks before the first drug administration (ascertained through inquiry).
* 7. Subjects who have used any mercaptopurine hydrate or thiopurine drugs within four weeks before the study (ascertained through inquiry).
* 8. Subjects who have heavily consumed, within 2 weeks prior to the first dose, or ingested within 48 hours prior to dosing, beverages containing caffeine or alcohol, or foods known to affect drug metabolism (such as chocolate, pitaya, mango, pomelo, carambola, guava, orange, grapefruit, or grapefruit products). (ascertained through inquiry)
* 9. Subjects who have undergone major surgical procedures (excluding diagnostic surgical procedures) within six months before the study , or those who plan to have surgery during the research period, or those who have undergone surgeries that, in the judgment of the researcher, can affect drug absorption, distribution, metabolism, and excretion (ascertained through inquiry).
* 10. Subjects who have received vaccination within three months before the study (ascertained through inquiry).
* 11. Subjects who have participated in any other clinical trial within 3 months prior to the current study. (Note: The end date is defined as the date of completion/exit from the previous clinical trial.) (ascertained through inquiry).
* 12. Subjects who have donated blood within three months before the study, or those whose total blood loss due to blood donation or other reasons has reached or exceeded 400 mL within six months (ascertained through inquiry).
* 13. Subjects who, on average, consumed more than 14 units of alcohol per week over the past year, or those unable to abstain from alcohol during the study period, or individuals with a breath alcohol test result greater than 0.0 mg/100 mL (ascertained through inquiry/examination).
* 14. Subjects who smoke more than 5 cigarettes per day on average within three months before the study, or those who cannot stop using any tobacco products during the study (ascertained through inquiry).
* 15. Subjects with a history of drug abuse (including the repeated and excessive use of various narcotic drugs and psychotropic substances for non-medical purposes) or positive results in drug abuse screening (including morphine, methamphetamine, ketamine, MDMA (3,4-methylenedioxymethamphetamine), cannabis (tetrahydrocannabinolic acid), etc.) within the past year (ascertained through inquiry and examination).
* 16. Subjects with a positive result in any item of the infectious disease examination during the screening period (including hepatitis B surface antigen, hepatitis C antibody, human immunodeficiency virus antibody, and treponema pallidum antibody) (examination).
* 17. Subjects who cannot tolerate venipuncture/indwelling needle or those with a history of fainting at the sight of needles or blood (ascertained through inquiry).
* 18. Subjects with difficult venous blood collection (ascertained through inquiry).
* 19. Subjects with lactose intolerance (ascertained through inquiry). 20. Subjects with special dietary requirements and who cannot accept the unified diet (ascertained through inquiry).
* 21. Subjects with dysphagia (ascertained through inquiry).
* 22. Other subjects are deemed unsuitable for participation by the researcher.
* 23. In addition to the above requirements, female subjects who meet the following conditions should also be excluded:
* a. Those who have used oral contraceptives within 30 days before the study (ascertained through inquiry).
* b. Those who have used long-acting estrogen or progesterone injections (including progesterone-containing intrauterine contraceptive devices) or implanted tablets within 6 months before the study (ascertained through inquiry).
* c. Those who have unprotected sexual intercourse with their partners within 14 days before the study (ascertained through inquiry).
* d. Those with a positive blood pregnancy test result (examination).
* e. Pregnant or lactating women (ascertained through inquiry).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Safety Assessment: Adverse Events (AEs) of single orally administered doses of F-02-2-Na in healthy adult subjects | From the start of the first dose to 72 hours after the last dose.
  Incidence, severity, and seriousness of adverse events (AEs) of single orally administered doses of F-02-2-Na in healthy adult subjects.
Safety Assessment: Proportion of subjects using Concomitant Medications during single orally administered doses of F-02-2-Na | From the start of the first dose to 72 hours after the last dose.
  Proportion of healthy adult Subjects Using Concomitant Medications during treatment with single orally administered doses of F-02-2-Na.
Safety Assessment: Proportion of subjects with Electrocardiogram (ECG) Findings following single orally administered doses of F-02-2-Na | From pre-dose (baseline) to 72 hours after the last dose.
  Proportion of healthy adult subjects with abnormal findings in electrocardiogram (ECG) parameters (including PR interval, QRS duration, QT/QTc interval, heart rate, and rhythm) following single orally administered doses of F-02-2-Na.
Proportion of subjects with abnormal hematology findings following single orally administered doses of F-02-2-Na | From pre-dose (baseline) to 72 hours after the last dose.
  Proportion of healthy adult subjects with clinically significant abnormalities in hematology parameters (e.g., hemoglobin, hematocrit, red blood cell count, white blood cell count with differential, platelet count) following single orally administered doses of F-02-2-Na.
Proportion of healthy subjects with abnormal coagulation findings following single orally administered doses of F-02-2-Na | From pre-dose (baseline) to 72 hours after the last dose.
  Proportion of healthy adult subjects with clinically significant abnormalities in coagulation parameters (e.g., PT, INR, aPTT) following F-02-2-Na.
Proportion of subjects with abnormal urinalysis findings following single orally administered doses of F-02-2-Na | From pre-dose (baseline) to 72 hours after the last dose.
  Proportion of healthy adult subjects with clinically significant abnormalities in urinalysis parameters (e.g., protein, glucose, blood, microscopic examination) following single orally administered doses of F-02-2-Na.
Proportion of subjects with abnormal clinical chemistry findings following single orally administered doses of F-02-2-Na | From pre-dose (baseline) to 72 hours after the last dose.
  Proportion of healthy adult subjects with clinically significant abnormalities in clinical chemistry parameters (e.g., sodium, potassium, chloride, calcium, ALT, AST, total bilirubin, alkaline phosphatase, creatinine, BUN, glucose) single orally administered doses of F-02-2-Na.
Proportion of subjects with abnormal renal morphology following single orally administered doses of F-02-2-Na | From pre-dose (baseline) to 72 hours post dose
  Proportion of healthy adult subjects with abnormal renal morphology as assessed by Renal Color Doppler Ultrasonography (Renal CDU) following single orally administered doses of F-02-2-Na.
Proportion of subjects with abnormal pelvicalyceal system findings following single orally administered doses of F-02-2-Na | From pre-dose (baseline) to 72 hours post dose
  Proportion of healthy adult subjects with abnormal pelvicalyceal system findings as assessed by Renal Color Doppler Ultrasonography (Renal CDU) following single orally administered doses of F-02-2-Na.
Proportion of subjects with abnormal renal vascular hemodynamics following single orally administered doses of F-02-2-Na | From pre-dose (baseline) to 72 hours post dose
  Proportion of healthy adult subjects with abnormal renal vascular hemodynamics as assessed by Renal CDU following single orally administered doses of F-02-2-Na.

SECONDARY OUTCOMES:
The effect of food on the pharmacokinetic Profile (Cmax) of F-02-2-Na in healthy adult subjects | From pre-dose (baseline) to 72 hours post dose
  To determine whether food intake affects key pharmacokinetic parameters: Cmax (maximum plasma concentration) of F-02-2-Na following single oral doses in healthy adult subjects.
The effect of food on the Pharmacokinetic Profile: Area Under the Concentration (AUC0-t) of F-02-2-Na in healthy Adult Subjects | From pre-dose (baseline) to 72 hours post dose
  To determine whether food intake affects key pharmacokinetic parameters: Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration (AUC0-t) of F-02-2-Na following single oral doses in healthy adult subjects.
The effect of food on the Pharmacokinetic Profile: Area Under the Concentration (AUC0-∞) of F-02-2-Na in healthy Adult Subjects | From pre-dose (baseline) to 72 hours post dose
  To determine whether food intake affects key Pharmacokinetic parameters: Area Under the Concentration-Time Curve from Time 0 to Extrapolated Infinity (AUC0-∞) of F-02-2-Na following single oral doses in healthy adult subjects.
The effect of food on the Pharmacokinetic Profile: Time to Maximum Plasma Concentration (Tmax) of F-02-2-Na in healthy Adult Subjects | From pre-dose (baseline) to 72 hours post dose
  To determine whether food intake affects key pharmacokinetic parameters: Time to reach maximum plasma concentration (Tmax) of F-02-2-Na following single oral doses in healthy adult subjects.
The effect of food on the Pharmacokinetic Profile: Terminal Elimination Half-Life (t1/2) of F-02-2-Na in Adult Subjects | From pre-dose (baseline) to 72 hours post dose
  To determine whether food intake affects key pharmacokinetic parameters: Terminal elimination half-life (t1/2) of F-02-2-Na following single oral doses in healthy adult subjects.
Absolute Change in Serum Uric Acid (sUA) Levels in healthy Adult Subjects After Single Oral Administrations of F-02-2-Na | From pre-dose (baseline) to 72 hours post dose
  To evaluate the absolute change in serum uric acid (sUA) levels in healthy adult subjects after single oral administrations of F-02-2-Na. The absolute change is calculated as the difference between sUA levels at each predefined time point and the baseline sUA level (absolute change = sUA level at predefined time point - baseline sUA level).
Percentage Change in Serum Uric Acid (sUA) Levels in healthy Adult Subjects After Single Oral Administrations of F-02-2-Na | From pre-dose (baseline) to 72 hours post dose
  To evaluate the percentage change in serum uric acid (sUA) levels in healthy adult subjects after single oral administrations of F-02-2-Na tablets. The percentage change is calculated relative to the baseline sUA level at each predefined time point (percentage change = [(sUA level at predefined time point - baseline sUA level)/baseline sUA level] × 100%).
Uric Acid Excretion (AeUR) in healthy Adult Subjects After Single Oral Administrations of F-02-2-Na | From pre-dose (baseline) to 72 hours post dose
  To evaluate the uric acid excretion (AeUR) in healthy adult subjects after single oral administrations of F-02-2-Na. AeUR is defined as the total amount of uric acid excreted in urine within a specified time period (e.g., 24 hours or predefined intervals after administration), reflecting the cumulative excretion capacity of uric acid.
Uric Acid Clearance Rate (CLUR) in healthy Adult Subjects After Single Oral Administrations of F-02-2-Na | From pre-dose (baseline) to 72 hours post dose
  To evaluate the uric acid clearance rate (CLUR) in healthy adult subjects after single oral administrations of F-02-2-Na. CLUR is calculated as the ratio of uric acid excretion rate to serum uric acid concentration (CLUR = AeUR / AUC_sUA), reflecting the efficiency of renal uric acid clearance, with the unit of volume per unit time (e.g., mL/min).
Area Under the Curve (AUC) of Serum Uric Acid (sUA) Dynamic Change Curve in healthy Adult Subjects After Single Oral Administrations of F-02-2-Na | From pre-dose (baseline) to 72 hours post dose
  To evaluate the area under the curve (AUC) of the serum uric acid (sUA) dynamic change curve in healthy adult subjects after single oral administrations of F-02-2-Na. AUC is calculated by integrating the sUA concentration-time curve over a predefined time period (e.g., AUC₀-t, AUC₀-∞), reflecting the total exposure level of sUA during the observation period, with the unit of concentration × time (e.g., μmol·h/L).
Total 24-Hour Uric Acid Excretion in healthy Adult Subjects After Single Oral Administrations of F-02-2-Na | From pre-dose (baseline) to 72 hours post dose
  To evaluate the total 24-hour uric acid excretion in healthy adult subjects after single oral administrations of F-02-2-Na. It is determined by collecting 24-hour urine samples, measuring the uric acid concentration in the urine, and calculating the total amount of uric acid excreted in 24 hours (Total 24-hour uric acid excretion = Urine uric acid concentration × 24-hour urine volume), with the unit of mass (e.g., mg/24h or mmol/24h).

CONTACTS AND LOCATIONS:
Overall Officials: Junyan Wu, MS, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Donghui Zheng, MM, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
This is a Phase I exploratory study, and the data involves core information related to drug development. Therefore, there are no current plans to share Individual Participant Data (IPD).

REFERENCES:
- [Background] Wang Z, Li X, Jin Y, Liu R, Di X, Zhou Y, Wang Y, Fan L, Chen Y, Wang Y, Zheng L. Safety, Efficacy, and Pharmacokinetics of HP501 in Healthy Volunteers and Hyperuricemic Patients: A Phase I/IIa Study. J Clin Endocrinol Metab. 2022 May 17;107(6):1667-1678. doi: 10.1210/clinem/dgac032. PMID 35106590
- [Background] Ding R, Chen L, Li X, Xiong T, Chen H, Hu X, Li Y, Zhou Y, Liu K, Wu J, Jiang F, Peng Q. A Phase I Study to Evaluate the Pharmacokinetic Drug-Drug Interaction of HP501, Febuxostat, and Colchicine in Male Chinese Patients with Hyperuricemia. Clin Drug Investig. 2023 Jun;43(6):401-411. doi: 10.1007/s40261-023-01274-7. Epub 2023 May 30. PMID 37248357
- [Background] Hall J, Gillen M, Yang X, Shen Z. Pharmacokinetics, Pharmacodynamics, and Tolerability of Concomitant Administration of Verinurad and Febuxostat in Healthy Male Volunteers. Clin Pharmacol Drug Dev. 2019 Feb;8(2):179-187. doi: 10.1002/cpdd.463. Epub 2018 Apr 24. PMID 29688628
- [Background] Lee HA, Yu KS, Park SI, Yoon S, Onohara M, Ahn Y, Lee H. URC102, a potent and selective inhibitor of hURAT1, reduced serum uric acid in healthy volunteers. Rheumatology (Oxford). 2019 Nov 1;58(11):1976-1984. doi: 10.1093/rheumatology/kez140. PMID 31056705